CLINICAL TRIAL: NCT05796505
Title: Addressing Vaccine Acceptance in Carceral Settings Through Community Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000035026; 1R01MD016853-01A1 (NIH)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Rapid cycle cluster randomized controlled trial (RCT). Randomization will occur at different levels, depending on the intervention that is being tested. Interviews: 14 key informant interviews will be conducted within each state correctional system that is identified as high performing (high vaccination rates for staff and incarcerated individuals). For rapid RCT: Pennsylvania Department Of Corrections operates 23 prisons which incarcerate approximately 35000 men and 1800 women. Every incarcerated individual in a PA prison is a potential candidate for the rapid RCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Participants receive standard interventions currently in use (treatment as usual).
- ADVANCE Steering Committee chosen interventions (Experimental): Interventions will be selected by the ADVANCE Steering Committee and will be rapidly deployed without additional effort on the part of front-line staff at four distinct levels: patient, provider, practice and prison level. Interventions will be tested one at a time in an iterative process. A participatory, assets-based framework will be used to identify acceptable and feasible strategies to improve vaccine acceptance. Each round of testing will include 1 month of preparation by the steering committee,12-week intervention period, and 2 months for analysis and rapid dissemination.
  Interventions: Behavioral: ADVANCE Steering Committee interventions

INTERVENTIONS:
Behavioral: ADVANCE Steering Committee interventions — Interventions will be selected by the ADVANCE Steering Committee and will be rapidly deployed without additional effort on the part of front-line staff at four distinct levels: patient, provider, practice and prison level. Interventions will be tested one at a time in an iterative process. A participatory, assets-based framework will be used to identify acceptable and feasible strategies to improve vaccine acceptance. Each round of testing will include 1 month of preparation by the steering committee,12-week intervention period, and 2 months for analysis and rapid dissemination.
  Arms: ADVANCE Steering Committee chosen interventions

SUMMARY:
The goal of this study is to reduce morbidity and mortality from COVID-19 amongst people who are detained in and work in correctional facilities. The overall objective is to identify feasible and effective interventions to improve vaccine uptake in correctional facilities and study the effectiveness of these interventions through rapid cycle, cluster randomized trials in the Pennsylvania prison system.

DETAILED DESCRIPTION:
Aim 1: To identify correctional system strategies to address COVID-19 and influenza vaccine acceptance amongst incarcerated people and correctional staff.

Aim 2: To select feasible strategies for a statewide correctional system at the patient-, provider-, practice- and prison-level to address COVID-19 and influenza vaccine uptake through a community engaged research approach.

Aim 3: To compare the effectiveness of interventions to address COVID-19 and influenza vaccine acceptance using a rapid cycle cluster randomized trial design in prison.

This study is highly innovative in its application of rapid cycle, cluster randomized trials in correctional systems to test the effectiveness of strategies identified using a community based participatory research approach. The results will serve as an evidence base for improving vaccine uptake that can be scaled nationally and adapted for other populations affected by the criminal legal system.

ELIGIBILITY:
Inclusion Criteria:

* All incarcerated people in the Pennsylvania DOC are included in the study population for these low risk interventions. In this each individual intervention, inclusion criteria will be based on where incarcerated people are housed and therefore what intervention they will be exposed to.

Exclusion Criteria:

* Exclusion criteria will likely include severe physical or mental illness as these individuals are often incarcerated in special units which will not be included in the study (i.e. medical units).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37122 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine acceptance rate | up to 12 weeks post intervention
  COVID-19 vaccine acceptance rate amongst incarcerated people and correctional staff assessed as the number of participants that receive a COVID-19 vaccine dose or complete the COVID-19 vaccine series by electronic health record (EHR) or self report. This will apply to anyone not fully up-to-date with the full immunization series, which is defined as inclusive of boosters.

SECONDARY OUTCOMES:
COVID-19 infections | up to 12 weeks post intervention
  Number of participants with COVID-19 infections by EHR or self report.
Hospitalization Rate | up to 12 weeks post intervention
  Total number of new admissions for COVID-19 infections by EHR or self report.
Deaths | up to 12 weeks
  Number of deaths from COVID-19 infections by EHR
Change in vaccination for other respiratory outbreaks | up to 12 weeks
  Change in vaccination rates for other respiratory outbreaks during winter season including influenza vaccine
Vaccine refusal rate | up to 12 weeks post intervention
  Vaccine refusal rate assessed by number of vaccines refused/total number fully vaccinated at start of the intervention
Vaccine acceptance rate | up to 12 weeks post intervention
  Vaccine acceptance rate assessed by number of vaccines administered/total number fully vaccinated at start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B Puglisi, MD, Principal Investigator — Yale University
Locations (1):
- Pennsylvannia Department of Corrections, Schwenksville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No